CLINICAL TRIAL: NCT05768113
Title: A Randomized, Double-blind, Multi-center Study to Evaluate the Efficacy and Safety of Ethyl Lauroyl Arginate Hydrochloride (LAEH) Formulation Versus a Matching Placebo Formulation
Brief Title: LAEH Formulation Nasal Spray to Reduce Viral Load
Status: Completed | Type: Observational
Sponsor: Salvacion USA Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SLV-CV19-SPRAY
Record Dates: First submitted 2023-01-06; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covixyl-V ELAH: No formal sample size calculation was performed. A total of 30 patients were enrolled and considered as sufficient sample size to compare the estimates of tests treatment with reference treatment
- Placebo: No formal sample size calculation was performed. A total of 30 patients were enrolled and considered as sufficient sample size to compare the estimates of tests treatment with reference treatment. This one is Placebo

SUMMARY:
The Covixyl-V LAEH Nasal Spray's safety and efficay is clinically tested for use in subjects with COVID-19 infection.

A randomized, double-blind, multi-center study is conducted to evaluate the efficacy and safety of ethyl lauroyl arginate hydrochloride (LAEH) formulation versus a matching placebo formulation administered as a nasal spray to reduce viral load from nasal area of subjects with coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
The primary endpoint for this study was the comparison of change in viral load in RT-PCR Test.

Proportion of COVID-19 infection-free subjects between the two treatment arms was followed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent or, by his or her legal/authorized representatives when the subject is not capable of giving consent, prior to initiation of any study procedures
2. Male or female of ≥18 years and ≤65 years of age (inclusive) at time of enrollment
3. Subjects with laboratory-confirmed diagnosis of COVID-19 at the time of screening (Day -3 to 0) using RT PCR method.
4. Subject with mild COVID-19 symptoms (e.g., fever, cough, sore throat, headache, muscle pain, nasal congestion, rhinorrhea, loss of smell and taste) but who did not have shortness of breath or dyspnea
5. Subjects who did not require hospitalization
6. Subjects with SpO2 levels ≥ 95%
7. Viral load by RT-PCR between 3.3 × 106 copies/mL to 6.6 × 106 copies/mL
8. Female subject who was not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile
9. Female subject of childbearing potential who had negative urine pregnancy test.

Exclusion Criteria:

1. Allergy to LAEH or any of the excipients of the formulation
2. History of allergies or flu within 30 days prior to the day of enrollment
3. Sensitivity to nostril skin or irritation or bleeding history within 30 days prior to the day of enrollment
4. Females who were breast-feeding, lactating, pregnant or intending to become pregnant
5. COVID-19 subjects with moderate, severe or critical illness or requiring intensive care or mechanical ventilation
6. History of severe respiratory disease and requirement for long-term oxygen therapy
7. Had received antibiotic/s, antiviral drug, and hormonal drugs within 30 days prior to the day of enrollment
8. Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator
9. Had received or had a plan to receive a SARS-CoV-2 vaccine during the study period
10. Participated in any interventional drug or medical device trials within 30 days prior to the day of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, 33 subjects were screened and 3 of them failed in screening tests. Total 30 subjects were enrolled in the study. Out of these 30 enrolled subjects, 15 subjects were randomized to Covixyl-V group and 15 subjects were randomized to placebo group
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Enumerating viral load using RT-PCR test. | 6days
  Comparison of change in viral load from baseline between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Amaya P Amaya, MD, Principal Investigator — 8485 Bird Road, Suite 303, Miami FL 33155
Locations (1):
- Global Clinical Trials, LLC,, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT05768113/Prot_SAP_000.pdf